CLINICAL TRIAL: NCT03178175
Title: Acupuncture for Management of Balance Impairment in Patients With Parkinson's Disease: A Single Blinded Randomised Controlled Study
Brief Title: Acupuncture for Management of Balance Impairment in Patients With Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study will be terminated due to poor patient recruitments.
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1051004
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease; Acupuncture
Keywords: Scalp acupuncture; Parkinson's disease; Balance
MeSH Terms: conditions — Parkinson Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture with "De Qi" (Experimental): all participants in this group will receive the standard procedure of acupuncture.
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): In this group, all participants will receive acupuncture needle insertion but not exact acupoint's location and depth.
  Interventions: Procedure: Needle Insertion

INTERVENTIONS:
Procedure: Acupuncture — In the acupuncture with "De Qi" group, using stainless tiny needles is inserted to the specific acupoints over the scalp (Si Shen Cong and Baihui) until the "De Qi" phenomenon occurs. The duration is about 30 minutes, and all patients will receive the procedure 16 times within 2 months.
  Arms: acupuncture with "De Qi"
Procedure: Needle Insertion — In the Sham acupuncture group, using stainless tiny needles is inserted to the specific acupoints over the scalp (Si Shen Cong and Baihui) but the needle doesn't reach the exact depth and "De Qi" phenomena doesn't occur. The duration is about 30 minutes, and all patients will receive this procedure 16 times within 2 months.
  Arms: Sham acupuncture

SUMMARY:
This plan is to evaluate the effectiveness of scalp acupuncture, a modern acupuncture technique specialized to neurological disorders, in managing motor function and body balance for PD patients. This is a randomized, controlled, single-blind clinical trial.

DETAILED DESCRIPTION:
BACKGROUND: Parkinson's disease (PD) is an age-related progressive neurodegenerative disease. The etiology and pathogenetic mechanisms that cause PD are still not fully understood. Scalp acupuncture (SA), a common treatment modality within complementary and alternative medicine, has been widely used for PD.

OBJECTIVE: To evaluate the effectiveness of scalp acupuncture, a modern acupuncture technique specialized to neurological disorders, in managing motor function and body balance for PD patients.

DESIGN: Randomized, controlled, single-blind clinical trial. SETTING: Department of Neurology, Chang Bing Show Chwan Memorial Hospital in Changhua County.

PARTICIPANTS: Patients with PD of grade 1 to 3 of Hoehn & Yahr (H&Y) scale (N = 26).

INTERVENTIONS: SA group (Si Shen Cong and Baihui) or control group. The techniques were administered by traditional chinese medicine trained in SA and evaluated at baseline and at 20 and 30 minutes.

MAIN OUTCOME MEASURE: Motor score subscale of Unified Parkinson's Disease Rating Scale (UPDRS) was used to measure the motor performances. Balance ability in each patient was assessed as follows: subjects were placed on a force platform (SPS, SYNAPSYS posturography system) to assess the displacement area from the centre of gravity, either with eyes open or closed, in a standing posture. The mini balance evaluation systems test (the mini-BESTest) was used to measure the performance of balance and walking speed. The test was repeated twice each in baseline period, SA period and post-SA period. The Mann-Whitney U test, Chi-square test, and Fisher's exact test were used to compare the baseline characteristics of the 2 groups. One-way repeated measures ANOVA was used to examine the differences among different time points (before, during, and after acupuncture treatment) within a group. Association between continuous variables was evaluated with Spearman's rank correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* age 50-75
* Meet the diagnostic criteria of Parkinson's disease: UK (United Kingdom) Parkinson's disease society brain bank clinical diagnostic criteria
* Disease severity of Hoehn-Yahr stage: stage I to III
* clinical condition stable, not adjusting medicine in recent 3 months
* no falling episode in recent 1 year
* live independently

Exclusion Criteria:

* already enrolled in another studies
* can't cooperate this evaluation examinations due to poor visual acuity, impaired cognitive function, musculoskeletal system disorder, or psychiatric illness
* any other condition would make participants not to cooperative this study
* can't tolerate acupuncture procedure

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Balance function evaluation | 15-20 minutes
  check participants' balance function by mini-BESTest (mini-Balance Evaluation Systems Test)

SECONDARY OUTCOMES:
Motor function evaluation | 15-20 minutes
  check participant's motor function by UPDRS (Unified Parkinson's Disease Rating Score)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsien Hung, M.D., Principal Investigator — Chang Bing Show Chang Memorial Hospital
Locations (1):
- Chang Bing Show Chwan Memorial Hospital, Chang-hua, Taiwan

IPD SHARING:
Plan to Share IPD: No